CLINICAL TRIAL: NCT00371852
Title: Safety Dermatological Evaluation of Topic Compatibility (Primary and Accumulated Dermical Irritability and Dermical Sensibility) of Dermacyd Wipes
Brief Title: Topic Compatibility Dermacyd Wipes - Lactoserum - Hygiene
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LACTO_L_01811
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Last update posted 2008-05-16 (Estimated); Status verified 2008-05

CONDITIONS: Hygiene
MeSH Terms: interventions — lactoserum

INTERVENTIONS:
Drug: lactoserum

SUMMARY:
The purpose of this study is to demonstrate the absence of irritation potential (primary dermic irritability and cumulated dermic irritability) and allergy (sensibilization) of the product Dermacyd wipes.

ELIGIBILITY:
Inclusion Criteria:

* Phototypes: I, II, III and IV;
* Integral skin test in the region;

Exclusion Criteria:

* Lactation or gestation
* Use of Anti-inflammatory and/or immune-suppression drugs
* Personnel history of atopy;
* History of sensibilization or irritation for topic products;
* Active cutaneous disease;
* Use of new drugs and/or cosmetics during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50
Dates: Start 2006-05

PRIMARY OUTCOMES:
Score evaluation of the cutaneous reaction, preconized by International Contact Dermatitis Research Group (ICDRG)

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-aventis, São Paulo, São Paulo, Brazil